CLINICAL TRIAL: NCT05333068
Title: COMBINEd Ischemia and Vulnerable Plaque Percutaneous INTERVENtion to Reduce Cardiovascular Events
Brief Title: COMBINE-INTERVENE: COMBINEd Ischemia and Vulnerable Plaque Percutaneous INTERVENtion to Reduce Cardiovascular Events
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diagram B.V. (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9357
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Multivessel Coronary Artery Disease; Ischemia; Vulnerable Plaque; Coronary Artery Disease
MeSH Terms: conditions — Ischemia; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MVD > 2 50% angiographic stenosis PCI revascularization strategy based FFR and OCT assessment (Experimental): MVD > 2 50% angiographic stenosis PCI revascularization strategy based FFR and OCT assessment
  Interventions: Procedure: PCI revascularization strategy based on combined FFR and OCT assessment
- MVD > 2 50% angiographic stenosis PCI revascularization strategy based FFR assessment (and sham OCT) (Sham Comparator): MVD > 2 50% angiographic stenosis PCI revascularization strategy based FFR assessment (and sham OCT)
  Interventions: Procedure: PCI revascularization strategy based FFR assessment

INTERVENTIONS:
Procedure: PCI revascularization strategy based on combined FFR and OCT assessment — PCI revascularization strategy based on combined FFR and OCT assessment All FFR ≤ 0.75 and Vulnerable plaque will be treated. VP defined as TCFA ( cap thickness ≤ 75 micron); Ruptured plaque; or Plaque erosion with > 70 % AS or MLA < 2.5 mm2.
  Arms: MVD > 2 50% angiographic stenosis PCI revascularization strategy based FFR and OCT assessment
Procedure: PCI revascularization strategy based FFR assessment — PCI revascularization strategy based FFR assessment (all lesions with FFR≤0.80 will be treated)
  Arms: MVD > 2 50% angiographic stenosis PCI revascularization strategy based FFR assessment (and sham OCT)

SUMMARY:
The COMBINE-INTERVENE Trial will investigate whether a PCI revascularization strategy based on combined FFR and OCT assessment is superior to a PCI revascularization strategy based on FFR-alone in patients with MVD with any presentation.

DETAILED DESCRIPTION:
The published COMBINE trial shows that patients carrying an OCT-detected thin-cap atheroma have a fivefold higher rate of the primary endpoint compared to patients without vulnerable lesion morphology, despite absence of ischemia. The most important finding of this trial is that not ischemia, but underlying lesion morphology could be the most important factor that predicts future adverse events. Together with the recently published ISCHEMIA trial, where ischemia guided revascularization failed to improve clinical outcomes compared to medical treatment, the COMBINE trial leads to a new way of thinking in interventional cardiology and also opens the door for new treatment strategies where a combined ischemic and morphologic assessment could lead to better clinical outcomes.

The COMBINE-INTERVENE Trial will investigate whether a PCI revascularization strategy based on combined FFR and OCT assessment is superior to a PCI revascularization strategy based on FFR-alone in patients with MVD with any presentation. The COMBINE-INTERVENE Trial is the first in line trial that will test focal percutaneous stenting for vulnerable plaque lesions independently from ischemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing PCI, aged 30-80 years with any clinical presentation
2. Angiographic criteria: presence of ≥ 2 de novo target lesions* located in 2 different native coronary arteries feasible for treatment with PCI (operator / Heart team decision)

Angiographic criteria target lesion* (all criteria I-IV should be applicable):

I. DS ≥ 50% on visual estimation II. de novo lesion located in native (non-grafted) vessel III. lesion reference diameter of ≥ 2.0 mm IV. Thrombolysis In Myocardial Infarction (TIMI) 3 flow in all vessels (with exclusion of culprit lesions if MI at presentation)

*Target lesions are either culprit MI lesions or lesions where FFR will be performed. Patients are eligible if they have ≥ 2 target lesions or one culprit and ≥ 1 target lesion.

Exclusion Criteria:

1. Patients with MVD requiring coronary artery bypass grafting (CABG) treatment (operator / local heart team decision)
2. Lesion located in a grafted segment or in a vein graft
3. In-stent restenosis lesions
4. Left main trifurcation
5. Left main lesion stand-alone (without other lesions)
6. Patients with severe tortuous lesions (where FFR and OCT is judged impossible or dangerous)
7. Chronic total occlusion
8. Spontaneous coronary dissection
9. Patients with severe valvular heart disease likely to require cardiac surgery within the next 2 years
10. Patients with left ventricle (LV) function less than 30%
11. Renal insufficiency (Glomerular Filtration Rate (GFR) < 29 ml/min/1.73m2; Kidney Disease Outcomes Quality Initiative (KDOQI) stage 4 and 5)
12. Life expectancy less than 3 years

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1222 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
cardiac death, any myocardial infarction (MI) or any clinically-driven revascularization at 24 months | 24 months
  cardiac death, any myocardial infarction (MI) or any clinically-driven revascularization at 24 months

SECONDARY OUTCOMES:
Cardiac death, any MI or any clinical-driven revascularization at 24 months excluding TLR events in all lesions with a FFR between 0.76-0.80 left untreated in the experimental arm | 24 months
  Cardiac death, any MI or any clinical-driven revascularization at 24 months excluding TLR events in all lesions with a FFR between 0.76-0.80 left untreated in the experimental arm
Cardiac death, any spontaneous MI or any clinically-driven revascularization at 24 months | 24 months
  Cardiac death, any spontaneous MI or any clinically-driven revascularization at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Elvin Kedhi, Prof.dr., Principal Investigator — Professor of Medicine McGill University; Director Intervention Cardiology, McGill University Health Center, Canada; Visiting Professor, Silesian Medical University Katowice, Poland
Locations (49):
- Monash Medical, Clayton, Australia
- Canada (3):
  - McGill University Health Centre, Montreal
  - Hamilton Health Sciences, Ontario
  - Niagara Health System - St. Catherines Site, Ontario
- Aarhus University Hospital, Aarhus, Denmark
- North-Estonia Medical Centre, Tallinn, Estonia
- France (2):
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Clinique Louis Pasteur, Nancy
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
- India (3):
  - Apex Heart Institute, Ahmedabad
  - Apollo Hospitals, Bangalore
  - Post Graduate Institute of Medical education and Research, Chandigarh
- Italy (2):
  - Humanitas Research Hospital, Milan
  - Policlinico Universitario Fondazione Agostino Gemelli, Rome
- Japan (2):
  - National University Corporation Institute of Science Tokyo, Bunkyō City
  - Yokohama City University Medical Center, Yokohama
- National Heart Institute, Kuala Lumpur, Malaysia
- Netherlands (4):
  - OLVG, Amsterdam
  - Albert Schweitzer Hospital, Dordrecht
  - Medisch Spectrum Twente, Enschede
  - Elisabeth-TweeSteden Hospital, Tilburg
- Wellington Hospital, Wellington, New Zealand
- Poland (6):
  - Medical University of Silesia, Katowice
  - Jagiellonian University; John Paul II Hospital, Krakow
  - University Hospital Krakow, Krakow
  - Miedziowe Centrum Zdrowia, Lubin
  - Warsaw Medical University, Warsaw
  - Regional Specialist Hospital, Wroclaw
- Romania (3):
  - C.C. Iliescu Institute of Cardiology Bucharest, Bucharest
  - Nicolae Stăncioiu Heart Institute, Cluj-Napoca
  - Clinic Hospital Targu Mures & S.C. Cardio Med SRL, Târgu Mureş
- Middle Slovak Institute of Cardiovascular Disease, Banská Bystrica, Slovakia
- Spain (9):
  - Hospital Bellvitge Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital de La Princesa, Madrid
  - Hospital Gregorio Marañón Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - University Hospital La Paz, Madrid
  - Marqués de Valdecilla University Hospital, Santander
  - Hospital La Fe Valencia, Valencia
- Sweden (4):
  - Linköping University, Linköping
  - Lund University, Lund
  - Universitetssjukhuset Örebro, Örebro
  - Danderyd Hospital, Stockholm
- Taiwan (3):
  - Far Eastern Memorial Hospital, New Taipei City
  - Cheng Hsin General Hospital, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Diagram B.V. — https://diagramresearch.com/trials/